CLINICAL TRIAL: NCT07040696
Title: Accuracy of the Venous Excess Ultrasound Score at Hospital Admission to Predict Acute Kidney Injury in Preeclampsia With Severe Features: A Prospective Observational Study
Brief Title: Accuracy of Venous Excess Ultrasound Score at Hospital Admission to Predict Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia, Cairo University
Other Study IDs: VEXUS score in preeclampsia
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Preeclampsia; Acute Kidney Injury
Keywords: preeclampsia; VEXUS score; AKI
MeSH Terms: conditions — Pre-Eclampsia; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preeclampsia with severe features: Features of severity will be defined according to American college of obstetric and gynacology guidelines
  Interventions: Device: Venous excess ultrasound score (VEXUS)

INTERVENTIONS:
Device: Venous excess ultrasound score (VEXUS) — Doppler examination of inferior vena cave, portal vein, hepatic vein, and intrarenal vein will be conducted by an experienced operator

SUMMARY:
To evaluate diagnostic accuracy of venous excess ultrasound score to predict acute kidney injury

DETAILED DESCRIPTION:
Preeclampsia is a common health problem during pregnancy. such condition may result in serious consequences including acute kidney injury. researchers of this study aim to evaluate the ability of venous excess ultrasound score at hospital admission to predict acute kidney injury in preeclampsia with severe features

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia with severe features

Exclusion Criteria:

* Patient refusal
* Preexisting renal impairment (defined as baseline serum creatinine > 1.3 mg/dl)
* Inability to obtain adequate Doppler views
* Renal transplantation
* Previous need for renal replacement therapy
* Known peripheral vascular disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Preeclampsia with severe features is defined according to the American College of Obstetricians and Gynecologists (ACOG)
Study Population: preeclampsia with severe features
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of VEXUS score at admission to predict acute kidney injury | within 48 hours of admission

SECONDARY OUTCOMES:
need for renal replacement therapy | at 28 days of admission
Cumulative fluid balance | within 48 hours of admission
In hospital mortality | At 28 days of admission

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may not be shared due to privacy regulations, ethical considerations

REFERENCES:
- [Background] Viana-Rojas JA, Argaiz E, Robles-Ledesma M, Arias-Mendoza A, Najera-Rojas NA, Alonso-Bringas AP, De Los Rios-Arce LF, Armenta-Rodriguez J, Gopar-Nieto R, Briseno-De la Cruz JL, Gonzalez-Pacheco H, Sierra-Lara Martinez D, Gonzalez-Salido J, Lopez-Gil S, Araiza-Garaygordobil D. Venous excess ultrasound score and acute kidney injury in patients with acute coronary syndrome. Eur Heart J Acute Cardiovasc Care. 2023 Jul 7;12(7):413-419. doi: 10.1093/ehjacc/zuad048. PMID 37154067
- [Background] Rola P, Miralles-Aguiar F, Argaiz E, Beaubien-Souligny W, Haycock K, Karimov T, Dinh VA, Spiegel R. Clinical applications of the venous excess ultrasound (VExUS) score: conceptual review and case series. Ultrasound J. 2021 Jun 19;13(1):32. doi: 10.1186/s13089-021-00232-8. PMID 34146184
- [Background] Naqvi R, Hossain N, Butt S, Bhellar Z, Fatima E, Imtiaz S, Moosa PG, Abbas K, Jafri SB, Khan S. Efficacy of multiple Biomarkers: NGAL, KIM1, Cystatin C and IL18 in predicting pregnancy related acute kidney injury. Pak J Med Sci. 2023 Jan-Feb;39(1):34-40. doi: 10.12669/pjms.39.1.6930. PMID 36694779
- [Background] Hassan M, Mayanja R, Ssalongo WGM, Robert N, Mark LH, Samson O, Muhindo R. Incidence and predictors of acute kidney injury among women with severe pre-eclampsia at Mbarara Regional Referral Hospital. BMC Nephrol. 2022 Nov 2;23(1):353. doi: 10.1186/s12882-022-02972-8. PMID 36324072